CLINICAL TRIAL: NCT05758779
Title: Coronary CT Screening of Patients With Familial Hypercholesterolemia - The Prevalence of Subclinical Atherosclerosis in Familial Hypercholesterolemia in the Region of Southern Denmark
Brief Title: The Danish Familial Hypercholesterolemia Organized Coronary Screening Trial
Acronym: DANFOCOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DANFOCOS
Record Dates: First submitted 2023-02-01; First posted 2023-03-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Familial Hypercholesterolemia; Atherosclerosis
Keywords: Familial Hypercholesterolemia; Subclinical Coronary Atherosclerosis; Coronary computerized tomography; Coronary arterial calcium score; Screening; Risc stratification
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary CT scan visualized for patient (Experimental): The patient is allowed to see the CT image of his/hers coronary vessels, including oral describtion of the findings.
  Interventions: Behavioral: Visualization of coronary Imaging and oral description
- Coronary CT scan NOT visualized for patient (No Intervention): The patient is not allowed to see the CT image of his/hers coronary vessels.

INTERVENTIONS:
Behavioral: Visualization of coronary Imaging and oral description — The participants is allowed to see their coronary CT scan including oral description. The study will test the effect on smoking habit and changes in LDL-C in one year.
  Arms: Coronary CT scan visualized for patient

SUMMARY:
Familial hypercholesterolemia (FH) is the most common inherited cause of atherosclerotic cardiovascular disease (ASCVD) with a prevalence of approximately one in 200 individuals, however only few of the estimated 30.000 patients with FH in Denmark has been diagnosed. FH is characterized by high levels of low-density lipoprotein cholesterol (LDL-C) and a high risk of premature ASCVD in particular coronary artery disease. The presence of atherosclerosis measured by cardiac computed tomography (CT) is a reliable predictor of future cardiovascular events and may help guide clinicians with regard to the lifestyle modifying therapies and lipid-lowering treatment. However, the prevalence and degree of coronary atherosclerosis in Danish FH patients without symptoms of ASCVD is unknown.

Therefore, the invetigators aimed to:

* Screen FH patients in a Danish setting for subclinical coronary atherosclerosis to improve lipid-lowering treatment and,
* Test if coronary CT screening can help to reach LDL-C therapy goals and reduce smoking.

This study will consist of a local cross sectional pilotstudy including 100 asymptomatic FH patients recruited from the lipid clinic at Odense University Hospital and hereafter a regional cross-sectional on approximately 600 asymptomatic FH patients in the Region of Southern Denmark recruited from the lipid clinics trough the national patient registry. In the pilot study, patients will undergo lipid analysis and non-contrast / contrast CT for description of coronary arterial calcium, and plaque morphology in this patient group. This will provide knowledge for planning the regional cross sectional study describing subclinical atherosclerosis in this population. Patients will furthermore be randomized to see their coronary CT scan or not. Mean LDL-C change and smoking status will be evaluated one year after.

The benefit of finding subclinical atherosclerotic disease with the possibility to improve lipid-lowering treatment for prevention of future premature ischemic heart disease is considered to outweigh the minor radiation exposure in this trial. If LDL-C is reduced significantly and smoking reduction is significant trough a simple intervention as showing the CT scan to the patient, this study can provide knowledge whether CT screening of this patient group should be considered in Denmark.

DETAILED DESCRIPTION:
1. Introduction:

   Familial hypercholesterolemia (FH) is the most common inherited cause of atherosclerotic cardiovascular disease (ASCVD) with a prevalence of 1/200. More than 30.000 patients in Denmark are expected to have FH, however, few of these patients is diagnosed.

   Patients with FH may have up to a 13-fold higher risk of coronary artery disease compared to the background population. However, FH can be treated with appropriate lipid-lowering treatment, and early initiation of lipid-lowering treatment may lower the risk of ASCVD to be comparable with individuals without FH. Early diagnosis and initiation of lifestyle modifying therapies and lipid-lowering treatment is of major importance to lower the risk of ASCVD in FH patients and their affected relatives. However, limited knowledge exist on whether risk stratification using objective measures of coronary artery atherosclerosis may be used to identify FH patients that require more intensive lipid-lowering treatment than others.

   FH should be suspected in individuals with severely elevated low-density lipoprotein - cholesterol (LDL-C) in, or in families with premature ASCVD. A diagnosis of FH is most often based on clinical scores such as the Simon Broome Criteria or the Dutch Lipid Clinical Network (DLCN) Criteria, which both include information on genetic testing for pathogenic FH mutations as an important part of making a definite diagnosis of FH.

   The lipid-lowering treatment in most FH patients include statins and ezetimibe. Proprotein-convertase-subtilisin/kexin-type 9 (PCSK9)-inhibitors are very potent and has been shown to reduce atherosclerotic plaques, but these agents are currently very expensive and their use in FH patients in the context of primary prevention is limited to patients with highly elevated LDL-C despite standard treatment.

   However FH remains under diagnosed, resulting in premature ASCVD and death. Thus, there is a need for optimized screening for ASCVD in asymptomatic FH patients for optimization in treatment.

   The Spanish SAFEHEART study was the first study to screen a larger population of patients with FH with coronary contrast and non-contrast CT scan for ASCVD. In this study 440 FH patients were included and screened with coronary CT and followed for a maximum of 3 years for development of cardiovascular disease. Interestingly, this study showed a significant prevalence of coronary atherosclerosis visualized by CT-scan, even in patients on lipid-lowering treatment, with 55% of the population with coronary calcium present. Coronary atherosclerosis is associated with increased risk of cardiovascular events, and the study concluded that coronary CT screening may be beneficial in risk stratification of asymptomatic FH patients, and that systematic screening potentially could benefit FH patients.

   However, whether CT screening for coronary atherosclerosis in asymptomatic FH patients has a potential in a Danish setting for risk stratification and optimizing in treatment remain unsettled. The recently published DANCAVAS 5 year outcome, found a benefit of CT-screening on all-cause mortality among men aged 65-69 years, and this support the rationale for screening younger patients in high-risk of ischemic heart disease. A minor study has been done with non-contrast coronary CT in Denmark including 88 FH patients in 2000, concluding that age adjusted coronary arterial calcium score (CACS) was strongly associated with ASCVD, however investigation of a larger population remains yet to be done.
2. Purpose:

   This study will by coronary CT screening investigate the prevalence of asymptomatic coronary atherosclerosis in patients with FH in the Region of Southern Denmark. The definition of subclinical coronary atherosclerosis will be finally settled through a pilot study describing coronary arterial calcium score (CACS), severity of stenosis, plaque composition and LDL-C in 100 patients with FH in different age groups.

   Furthermore participants will be randomized to see their coronary imaging at screening. Change in LDL-C and smoking status one year after screening will be evaluated as an indicator for optimized treatment.

   Finally, the investigators will screen for subjects beeing candidates for a future interventional study with intensified lipid lowering treatment with PCSK9-inhibitors.

   The investigators hypothesize that approximately 50% of the FH patients has subclinical atherosclerosis before the age of 50, and that coronary CT screening can be used for optimizing lipid-lowering treatment by stratifying FH patient according to presence of subclinical coronary atherosclerosis and adjusting LDL-C treatment targets. In addition, the investigators hypothesize that visualization of the coronary arteries for the patient is associated with a reduction in LDL-C and a reduction in smoking one year after screening.
3. Method:

   3.1 Design: The project include a cross-sectional pilot study that will be conducted at the Department of Cardiology at Odense University Hospital and a larger regional cross-sectional study, in cooperation with the departments of cardiology in the Region of Southern Denmark. Furthermore the study will include an imbeded Randomized Controlled Trial (RCT).

   3.2 Intervention: This is primary a cross sectional study screening asymptomatic patients with FH with coronary CT, describing the prevalence of subclinical atherosclerosis. Coronary CT scan will be performed according to the local guidelines for optimal imaging quality, Image analysis will be done using standard software for CACS analysis (Synovia, Siemens Healthineers solution, Forcheim Tyskland) and Autoplaq software (Cedars Sinai Medical Center, LA, California, USA).

   The study will include an imbeded RCT randomizing the patients to see or not see their coronary CT image, evaluating effect on cholesterol and smoking status. Questionary will be completed before CT-scanning and one year after CT scanning.

   3.2.1 Pilot study Initially a pilotstudy on 100 patients will be conducted at the Department of Cardiology at Odense University Hospital. Eligible patients will be identified at first contact or during follow-up in the lipid clinic. The eligible patients will be invited to participation in the trial by mail/letter containing information regarding the trial. If he/she is willing to participate in the study, informed consent is obtained at first visit and echocardiography, ultrasound of femoral and carotid arteries, and ECG will be performed and blood samples (lipidprofile, Hba1c, TSH, liver and kidney parameters) will be collected prior to coronary CT with and without contrast. The investigators aim to recruit patients evenly distributed on age and sex from 20-70 years.

   The purpose of the pilot study is to investigate the prevalence of coronary atherosclerosis in asymptomatic men and women in different age groups, providing knowledge for planning the regional cross sectional study.

   3.2.2 Regional cross-sectional study In the regional cross-sectional study, eligible patients with a diagnosis of FH will be identified through the National Patients Registry and in cooperation with the local lipid clinics. The investigators estimate that approximately 1000 will be eligible and that 600 will participate in the study. Eligible patients will be invited to participate in the trial at ambulatory contacts or by mail/letter containing information regarding the trial. Age group for invitation to the study will be settled according to findings from the pilot study, probably 30-70 years. If he/she is willing to participate in the study, informed consent will be obtained at first visit and echocardiography, ultrasound of femoral and carotid arteries, and ECG will be performed and blood samples (lipidprofile, Hba1c, TSH, liver and kidney parameters) will be collected prior to coronary CT.

   3.2.3 Imbedded RCT. 200 patients from the regional cross sectional study will be randomized to see or not see their coronary CT image. Follow up will be after one year, measuring LDL-C and evaluating smoking status by a survey. Outcome will be differences in LDL-C and probability of being a smoker, defined as odds ratio (OR) for being a smoker between the two groups.

   3.3 Sample size: The aim is to include 400 patients in a future pharmacological interventional study. Therefore the investigators aim to include 600 patients in the regional cross-sectional study taking account for exclusion/dropout of 25 % in the pharmacological interventional study.

   3.4 Randomisation In both the pilot study and the regional cross -sectional study, patients will be randomized to seeing their coronary CT image or not. LDL-C levels and smoking status will be evaluated after one year. The investigator analyzing endpoints will be blinded to whether the patients has seen there CT or not.

   3.5 Statistical analyses The pilot study will describe median CACS, plaque composition (proportion of soft versus calcified plaques), severity of stenosis and LDL-C levels.

   Statistical analysis on LDL-C change and smoking status one year after coronary CT screening and randomization to either seeing the coronary imaging or not will be performed by STATA.

   3.5.1 Numerical outcomes: For change in LDL-C levels and number of cigarettes per day after one year, the difference in means between the group seeing the coronary imaging and the group not seeing the coronary imaging will be calculated by Students T-test.

   3.5.2 Binary outcomes: For smoking status one year after randomization to seeing the coronary imaging or not, the probability for being a smoker, defined as odds ratio (OR) for being a smoker will be calculated by chi squared test.
4. Ethics:

   The average dose of one non-contrast cardiac CT scan is 1 mSv and the average dose of an additional contrast cardiac CT scan is 3 mSv.

   The 100 participants in the DANFOCOS pilot study will therefore receive 4 mSv, corresponding to one contrast and one non contrast cardiac CT scan.

   For comparison, the annual background radiation dose in Denmark is 3 mSv, and the average annual limit for radiation workers is 20 mSv. Overall the benefits of finding premature atherosclerotic disease with the possibility to improve treatment is considered to outweigh the radiation dose.
5. Organization:

   This Project is initiated from the cardiological department at Odense University Hospital as part of a PhD program with MD. Jakob Knold. The project will be associated with the Clinical Institute at University of Southern Denmark.

   The Steering Commitee will consist of main supervisor Associated Professor Finn Lund Henriksen (PI, Department of Cardiology OUH). Professor Axel Diederichsen (Department of Cardiology OUH), Associated Professor Kristian Altern Øvrehus (Department of Cardiology OUH), PhD Christian Sørensen Bork (Department of Cardiology AAUH). MD. Jakob Knold (Department of Cardiology OUH). The data registration will be performed via REDCap with logging and secure storage directly on a server under Odense Patient Data Explorative Network (OPEN), Region of Southern Denmark.
6. Economi and Funding Private and public foundations are sought for funding. The investigators has no economical affiliation or conflicts of interest.
7. Perspectives This study will be the largest screening of asymptomatic FH patients with coronary CT in a Danish setting and test if visualization of the coronary arteries for the patient has an effect on LDL-C levels and smoking status after one year. The study will identify patients with asymptomatic coronary atherosclerosis which require a lower LDL-C target than patients without coronary atherosclerosis and thereby elucidate whether coronary CT screening of FH patients can improve treatment of this patient group in Denmark. The study will identify eligible subjects for a future interventional study with intensified lipid lowering treatment (PCSK9-inhibitors), which could have implications for the current guideline regarding PCSK9-inhibitors, improving the treatment of FH patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with genetically or clinically FH (DLCN score > 6) between the age of 20 and 70 are eligible patients in DANFOCOS.

Exclusion Criteria:

* History of ASCVD defined as myocardialinfarction, procedural revascularisation, CABG and/or objective evidence if ischaemia (exercise stress test, stress echocardiography, myocardial perfusion scintigraphy, stress cardiac magnetic resonance, coronary angiography, cardiac CT), angina pectoris, ischaemic stroke or a medically (aspirin, clopidogrel, persantin) treated transitory ischaemic attack, and symptomatic peripheral vascular disease with ankle-brachial index below 0.9 or procedural revascularisation.
* Current Pregnancy or planning pregnancy (due to radiation issues)
* eGFR < 60 ml/min/1,73 m2 (due to CT-contrast)
* Prior allergic reaction to CT-contrast.
* PCSK9-inhibitor treatment
* Life expectancy < 5 years.
* Secondary dyslipidemia

  * Dysregulated diabetes
  * Dysregulated hypothyreosis TSH > 4,0 IU/L.
  * Combined hyperlipidemia: TG > 4 mmol/L
  * Nefrotic syndrome: proteinuria > 3 g/L and s-albumin < 30 g/l
  * History of primary billiary cirrhosis
  * Low-carb-high-fat diet.
  * Pharmacological induced dyslipidemia

Findings on Coronary CT leads to exclusion

* Three vessels disease
* Left main coronary artery stenosis
* Proximal left anterior descending coronary artery stenosis
* Proximal right coronary artery stenosis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Coronary arterial calcium score (CACS) | 18 months
  Mean CACS of the population
CACS | 18 months
  Median CACS of the population
Plaque composition | 18 months
  proportion of soft and calcified plaques
Plaque volume (mean) | 18 months
  Mean size of plaques described in mm.
Plaque volume (median) | 18 months
  Median size of plaques described in mm.
Severity of stenosis (number of stenosis) | 18 months
  Percentage of vessel lumen compromised by plaque described as number of minor, moderate and severe stenosis.
Severity of stenosis (proportion of stenosis) | 18 months
  Percentage of vessel lumen compromised by plaque described as proportion of minor, moderate and severe stenosis.

SECONDARY OUTCOMES:
Change in LDL-C levels. | 12 months
  Mean change in LDL-C levels one year after randomization to see coronary imaging. Difference in mean between the two groups
Change in smoking status | 12 months
  Odds ratio for being af smoker one year after randomization to see or not see your coronary imaging
Change in mean consumption cigarettes per day | 12 months
  Mean change in number of smoked cigarettes per day, one year after randomization to see coronary imaging. Difference in mean between the two groups
Prevalence of femoral and carotid plaques | 18 months
  Prevalence of femoral and carotid plaques visualized by ultrasound, described as proportion of plaques in the population.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Lund Henriksen, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levenson AE, de Ferranti SD. Familial Hypercholesterolemia. In: Feingold KR, Anawalt B, Boyce A, Chrousos G, de Herder WW, Dhatariya K, et al., editors. Endotext. South Dartmouth (MA)2000
- [Background] Bundgaard H SMea. Regionernes klinisk kvalitetsdatabase. Familiær hyperkolesterolæmi databasen. 2020 [Available from: https://www.rkkp.dk/kvalitetsdatabaser/databaser/databasen-for-familiaer-hyperkolesterolaemi/
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Rosso A, Pitini E, D'Andrea E, Massimi A, De Vito C, Marzuillo C, Villari P. The Cost-effectiveness of Genetic Screening for Familial Hypercholesterolemia: a Systematic Review. Ann Ig. 2017 Sep-Oct;29(5):464-480. doi: 10.7416/ai.2017.2178. PMID 28715059
- [Background] Sturm AC, Knowles JW, Gidding SS, Ahmad ZS, Ahmed CD, Ballantyne CM, Baum SJ, Bourbon M, Carrie A, Cuchel M, de Ferranti SD, Defesche JC, Freiberger T, Hershberger RE, Hovingh GK, Karayan L, Kastelein JJP, Kindt I, Lane SR, Leigh SE, Linton MF, Mata P, Neal WA, Nordestgaard BG, Santos RD, Harada-Shiba M, Sijbrands EJ, Stitziel NO, Yamashita S, Wilemon KA, Ledbetter DH, Rader DJ; Convened by the Familial Hypercholesterolemia Foundation. Clinical Genetic Testing for Familial Hypercholesterolemia: JACC Scientific Expert Panel. J Am Coll Cardiol. 2018 Aug 7;72(6):662-680. doi: 10.1016/j.jacc.2018.05.044. PMID 30071997
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Raal FJ, Hovingh GK, Catapano AL. Familial hypercholesterolemia treatments: Guidelines and new therapies. Atherosclerosis. 2018 Oct;277:483-492. doi: 10.1016/j.atherosclerosis.2018.06.859. PMID 30270089
- [Background] Hedegaard BS. A danish nationwide study og individuals suspected of FH referred from general practice to lipid clinics: Clinical characteristics, plasma lpipoprotein(A) and final diagnosis. Atherosclerosis. 2021.
- [Background] Schmidt EB, Hedegaard BS, Retterstol K. Familial hypercholesterolaemia: history, diagnosis, screening, management and challenges. Heart. 2020 Dec;106(24):1940-1946. doi: 10.1136/heartjnl-2019-316276. Epub 2020 Sep 15. No abstract available. PMID 32933999
- [Background] Perez de Isla L, Alonso R, Muniz-Grijalvo O, Diaz-Diaz JL, Zambon D, Miramontes JP, Fuentes F, Gomez de Diego JJ, Gonzalez-Estrada A, Mata N, Saltijeral A, Barreiro M, Tomas M, de Andres R, Argueso R, Serrano Gotarredona MP, Navarro Herrero S, Perea Palazon RJ, de Caralt TM, Suarez de Centi LA, Zhilina S, Espejo Perez S, Padro T, Mata P; SAFEHEART investigators. Coronary computed tomographic angiography findings and their therapeutic implications in asymptomatic patients with familial hypercholesterolemia. Lessons from the SAFEHEART study. J Clin Lipidol. 2018 Jul-Aug;12(4):948-957. doi: 10.1016/j.jacl.2018.04.003. Epub 2018 Apr 17. PMID 29753733
- [Background] Luirink IK, Kuipers IM, Hutten BA, Planken RN, Backx APCM, Groothoff JW, Wiegman A. Coronary computed tomography angiography and echocardiography in children with homozygous familial hypercholesterolemia. Atherosclerosis. 2019 Jun;285:87-92. doi: 10.1016/j.atherosclerosis.2019.04.219. Epub 2019 Apr 11. PMID 31048103
- [Background] Lindholt JS, Sogaard R, Rasmussen LM, Mejldal A, Lambrechtsen J, Steffensen FH, Frost L, Egstrup K, Urbonaviciene G, Busk M, Diederichsen ACP. Five-Year Outcomes of the Danish Cardiovascular Screening (DANCAVAS) Trial. N Engl J Med. 2022 Oct 13;387(15):1385-1394. doi: 10.1056/NEJMoa2208681. Epub 2022 Aug 27. PMID 36027560
- [Background] Jensen JM, Gerdes LU, Jensen HK, Christiansen TM, Brorholt-Petersen JU, Faergeman O. Association of coronary heart disease with age-adjusted aortocoronary calcification in patients with familial hypercholesterolaemia. J Intern Med. 2000 Apr;247(4):479-84. doi: 10.1046/j.1365-2796.2000.00630.x. PMID 10792562
- [Background] Wang W, Yang L, Wang S, Wang Q, Xu L. An automated quantification method for the Agatston coronary artery calcium score on coronary computed tomography angiography. Quant Imaging Med Surg. 2022 Mar;12(3):1787-1799. doi: 10.21037/qims-21-775. PMID 35284280
- [Background] Romanens M, Mortensen MB, Sudano I, Szucs T, Adams A. Extensive carotid atherosclerosis and the diagnostic accuracy of coronary risk calculators. Prev Med Rep. 2017 Mar 14;6:182-186. doi: 10.1016/j.pmedr.2017.03.006. eCollection 2017 Jun. PMID 28352516
- [Background] Preston DL, Ron E, Tokuoka S, Funamoto S, Nishi N, Soda M, Mabuchi K, Kodama K. Solid cancer incidence in atomic bomb survivors: 1958-1998. Radiat Res. 2007 Jul;168(1):1-64. doi: 10.1667/RR0763.1. PMID 17722996
- [Background] Einstein AJ, Knuuti J. Cardiac imaging: does radiation matter? Eur Heart J. 2012 Mar;33(5):573-8. doi: 10.1093/eurheartj/ehr281. Epub 2011 Aug 9. PMID 21828062